CLINICAL TRIAL: NCT00544128
Title: A Randomized, Open Label, Multicenter Study Comparing the Safety and Efficacy of Once Daily Regimen Containing Epzicom or Truvada Combined With Ritonavir Boosted Atazanavir as Initial Therapy for HIV-1 Infection (ET Study)
Brief Title: Comparison of Epzicom and Truvada for the Initial Once Daily HIV Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Medical Center of Japan (Other Government)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Principal Investigator, Shinichi Oka, M.D., Shinichi Oka, Director general, AIDS Clinical Center, International Medical Center of Japan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMCJ-H19-466; ET001
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: HIV; initial therapy; once daily; randomized trial; non inferiority; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Lamivudine; abacavir; Ritonavir; Atazanavir Sulfate; Emtricitabine; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epzicom Arm (Active Comparator): Patients are treated with Epzicom (lamivudine 300mg and abacavir 600mg) combined with ritonavir 100mg boosted atazanavir 300mg
  Interventions: Drug: lamivudine, abacavir , ritonavir, atazanavir
- Truvada Arm (Active Comparator): Patients are treated with Truvada (emtricitabine 200mg and tenofovir 300mg) combined with ritonavir 100mg boosted atazanavir 300mg
  Interventions: Drug: emtricitabine, tenofovir, ritonavir, atazanavir

INTERVENTIONS:
Drug: lamivudine, abacavir , ritonavir, atazanavir — Patients are treated with Epzicom (lamivudine 300mg and abacavir 600mg) combined with ritonavir 100mg boosted atazanavir 300mg
  Arms: Epzicom Arm
Drug: emtricitabine, tenofovir, ritonavir, atazanavir — Patients are treated with Truvada (emtricitabine 200mg and tenofovir 300mg) combined with ritonavir 100mg boosted atazanavir 300mg.
  Arms: Truvada Arm

SUMMARY:
A non-inferiority randomized control trial in treatment naïve HIV patients to compare virologic effect of two backbone regimens with Epzicom (lamivudine and abacavir) and Truvada (emtricitabine and tenofovir). Both arms are treated with fixed combination of ritonavir boosted atazanavir as key drugs.

DETAILED DESCRIPTION:
In treatment naïve HIV-1-infected patients, once daily combination antiretroviral therapy containing ritonavir boosted atazanavir combined with Epzicom will offer non inferior antiretroviral efficacy compared to ritonavir boosted atazanavir combined with Truvada. This non inferiority hypothesis is studied by a randomized, open label, multicenter trial over 48 weeks as the primary endpoint and long term safety of both arms are followed for 144 weeks.

The primary endpoint is the antiretroviral effect over 48 weeks.

The secondary endpoints are;

1. The immunologic effects from baseline at the 48th and 144th week
2. Reasons of treatment failure by 144th week
3. Adverse events and their rate of incidence by 144th week
4. Serum concentration of tenofovir in selected patients
5. Serum concentration of atazanavir in selected patients
6. Renal complication in tenofovir arm

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV infection,
* Antiretroviral initiation is recommended by current clinical guidelines,
* Treatment naïve,
* Age over 20 years old Japanese,
* Able to obtain written informed consent

Exclusion Criteria:

* Current malabsorption condition,
* Prior use of lamivudine for hepatitis B treatment,
* Positive serology of Hepatitis B surface antigen,
* Patients who have following abnormal laboratory results within 6 weeks prior enrollment;

  1. alanine aminotransferase is more than 2.5 times higher of upper normal limit
  2. estimated glomerular filtration rate is less than 60ml/min by Cockcroft-Gault equation
  3. serum phosphate level is less than 2.0mg/dl
* Patients with hemophilia, diabetes mellitus which require pharmacological treatment, congestive heart failure, cardiomyopathy or other serious medical condition
* Patients in pregnancy or breat feeding
* Patients who are taking medications contraindicated combine use of study medicine
* Patients whose primary care physicians consider inadequate to be enroll the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2007-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
antiretroviral effect over 48 weeks | 48 weeks

SECONDARY OUTCOMES:
The immunologic effects from baseline at the 48th and 144th week | 144 weeks
Reasons of treatment failure by 144th week | 144 weeks
Adverse events and their rate of incidence by 144th week | 144 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shinichi Oka, MD, Study Chair — International Medical Center of Japan
Locations (1):
- International Medical Center of Japan, Shinjuku, Tokyo, Japan

REFERENCES:
- [Result] Nishijima T, Takano M, Ishisaka M, Komatsu H, Gatanaga H, Kikuchi Y, Endo T, Horiba M, Kaneda S, Uchiumi H, Koibuchi T, Naito T, Yoshida M, Tachikawa N, Ueda M, Yokomaku Y, Fujii T, Higasa S, Takada K, Yamamoto M, Matsushita S, Tateyama M, Tanabe Y, Mitsuya H, Oka S; Epzicom-Truvada study team. Abacavir/lamivudine versus tenofovir/emtricitabine with atazanavir/ritonavir for treatment-naive Japanese patients with HIV-1 infection: a randomized multicenter trial. Intern Med. 2013;52(7):735-44. doi: 10.2169/internalmedicine.52.9155. Epub 2013 Apr 1. PMID 23545667